CLINICAL TRIAL: NCT00386061
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Fixed-Dose, Multicenter Study of Weight-Reducing Effect and Safety of SR141716 in Obese Patients With or Without Comorbidities (RIO-Europe)
Brief Title: Rimonabant in Obesity Over a 2-Year Duration (RIO-Europe)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sanofi (Industry)
Responsible Party: ICD Study Director, sanofi-aventis
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EFC4733
Record Dates: First submitted 2006-10-10; First posted 2006-10-11 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Obesity
Keywords: Obesity; risk factors
MeSH Terms: conditions — Obesity | interventions — Rimonabant

STUDY DESIGN:
Who Masked: Participant, Investigator

INTERVENTIONS:
Drug: rimonabant (SR141716)

SUMMARY:
The primary objective was to assess the effect of SR141716 on weight loss and weight maintenance over a period of one year when prescribed with a hypocaloric diet in obese patients with or without comorbidities.

The main secondary objectives were to assess the effect of SR141716 on lipid parameters (HDL-C, TG), glucose tolerance status, the rate of patients with metabolic syndrome, waist circumference, glycemic parameters.

ELIGIBILITY:
Inclusion Criteria:

* body mass index (BMI) e30 kg/m2 in patients with or without comorbidities, or BMI >27 kg/m2 in patients with treated or untreated hypertension and/or treated or untreated dyslipidemia.
* stable body weight (variation <5 kg within 3 months prior to screening visit);

Exclusion Criteria:

* History of very low-calorie diet within 6 months prior to screening visit; or history of surgical procedures for body weight loss (eg, stomach stapling, bypass);
* Presence of any clinically significant psychiatric , neurological or endocrine disease
* Presence of treated or untreated type 1 or type 2 diabetes);
* SBP >165 mmHg and/or DBP >105 mmHg on 2 consecutive visits from the screening to the inclusion visit;
* History of myocardial infarction or unstable angina pectoris within 6 months prior to screening visit; and history of stroke within 6 months prior to screening visit;
* Administration of anti-obesity drugs or other drugs for body weight reduction within 3 months prior to screening visit;

The investigator will evaluate whether there are other reasons why a patient may not participate.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1507 (Actual)
Dates: Start 2001-10; Primary Completion 2004-06 (Actual); Study Completion 2004-06 (Actual)

PRIMARY OUTCOMES:
change in body weight from baseline to 1 year.

SECONDARY OUTCOMES:
HDL-C and TG from baseline to 1 year; ·patients (%) with improvement of glucose tolerance, patients (%) with NCEP-ATPIII metabolic syndrome at 1 year.

CONTACTS AND LOCATIONS:
Overall Officials: ICD CSD, Study Director — Sanofi
Locations (7):
- Sanofi-Aventis, Bridgewater, New Jersey, United States
- Sanofi-Aventis, Brussels, Belgium
- Sanofi-Aventis, Helsinki, Finland
- Sanofi-Aventis, Paris, France
- Sanofi-Aventis, Berlin, Germany
- Sanofi-Aventis, Gouda, Netherlands
- Sanofi-Aventis, Bromma, Sweden

REFERENCES:
- [Result] Van Gaal LF, Rissanen AM, Scheen AJ, Ziegler O, Rossner S; RIO-Europe Study Group. Effects of the cannabinoid-1 receptor blocker rimonabant on weight reduction and cardiovascular risk factors in overweight patients: 1-year experience from the RIO-Europe study. Lancet. 2005 Apr 16-22;365(9468):1389-97. doi: 10.1016/S0140-6736(05)66374-X. PMID 15836887
- [Derived] Van Gaal LF, Scheen AJ, Rissanen AM, Rossner S, Hanotin C, Ziegler O; RIO-Europe Study Group. Long-term effect of CB1 blockade with rimonabant on cardiometabolic risk factors: two year results from the RIO-Europe Study. Eur Heart J. 2008 Jul;29(14):1761-71. doi: 10.1093/eurheartj/ehn076. Epub 2008 Apr 15. PMID 18417461